CLINICAL TRIAL: NCT05913336
Title: Evaluating the Efficacy and Safety of Remimazolam Tosilate for Injection for Prolonged Mechanical Ventilation Sedation in the Intensive Care Unit (ICU) - A Non-randomized, Multicenter, Single-arm, Open-label, Proof-of-concept, Phase I/II Clinical Trial
Brief Title: A Study of Remimazolam Tosilate for Prolonged Sedation in the ICU
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HR7056-206
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Sedation in the ICU

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remimazolam Tosilate (Experimental): IV of Remimazolam Tosilate
  Interventions: Drug: Remimazolam Tosilate

INTERVENTIONS:
Drug: Remimazolam Tosilate — Loading dose: 0.08mg/kg , Maintenance dose: IV remimazolam tosilate, dose range 0-2.0mg/kg/h, increment or decrement of 0.1-0.2mg/kg/h

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Remimazolam Tosilate for Injection for prolonged sedation(≥72h) during mechanical ventilation in the ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their guardians are able to provide a written informed consent
2. Subjects have been treated with endotracheal intubation and mechanical ventilation, and is expected to receive sedation after randomization. The target level and duration of sedation meet the criteria
3. Age ≥ 18 and ≤ 80 years, male or female
4. Body mass index (BMI) > 18 and < 30 kg/m2

Exclusion Criteria:

1. participants (other than in endotracheal intubation) who are expected to require neuro-muscle blockers during sedation；
2. Suffering from mental disorders (such as schizophrenia, depression, etc.) and cognitive dysfunction;
3. Organ failure during screening period；
4. Subjects who were receiving dialysis during the screening period or who were expected to require dialysis treatment during the study period;
5. History of epilepsy or status epilepticus;
6. Subjects with a history of drug abuse；
7. Myasthenia gravis or a history of myasthenia gravis;
8. severe arrhythmias or heart disease;
9. Subjects after neurosurgery operation；
10. participants who did not require continuous sedation during mechanical ventilation for endotracheal intubation;
11. Abnormal values of the laboratory examination
12. Subjects who required vasopressor medication to maintain normotensive blood pressure during the screening period (excluding subjects who used vasopressor medication only during surgery);
13. Allergic to relevant drugs ingredient or component;
14. Pregnant or nursing women;
15. Subjects who has participated in clinical trials of other interventions recently;
16. Other conditions deemed unsuitable to be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-27 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Rate of sedation success, sedation success is defined as the percentage of time maintaining target sedation in the entire drug administering time ≥ 70% without rescue sedation. | within 72 hours after administration of research drug

SECONDARY OUTCOMES:
Percentage of time maintaining target sedation in the entire drug administering time. | within 72 hours after administration of research drug
Percentage of subjects receiving rescue sedation and the average dosage of rescue sedation | within 72 hours after administration of research drug
Percentage of subjects receiving rescue analgesia and the average dosage of rescue analgesia | within 72 hours after administration of research drug
Wake-up time. | after stopping the research drug
Evaluation of nursing difficulty. | follow-up period (approx. 5-10 minutes)
Mechanical ventilation time. | at the time of extubation

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou, China

IPD SHARING:
Plan to Share IPD: Undecided